CLINICAL TRIAL: NCT00500214
Title: Ilioinguinal Nerve Excision in Open Mesh Repair of Inguinal Hernia,a Randomized Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Ilioinguinal nerve excision
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2007-07-12 (Estimated); Status verified 2007-07

CONDITIONS: Postoperative Pain; Postoperative Hyposthesia
Keywords: inguinal hernia; herniorrhaphy; mesh repair; ilioinguinal neurectomy; postoperative pain in cases and controls during one year.; postoperative hyposthesia in cases and controls during one year.
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: elective ilioinguinal nerve excision

SUMMARY:
this study was designed to evaluate the effect of routine excision of the ilioinguinal nerve in an attempt to decrease the incidence of chronic inguinodynia in patients who undergo open anterior hernia mesh repair.

DETAILED DESCRIPTION:
As chronic pain is the 2nd most common complication following open hernia repairs and it causes limitations and dysfunctions for the patients and also according to some previous studies elective ilioinguinal neurectomy could result in less postoperative pain,we decided to perform a randomized double blind clinical trial.The primary goal of this study was evaluation of the effect of this type of neurectomy on postoperative pain and hyposthesia.

ELIGIBILITY:
Inclusion Criteria:

* having an age of over 18 years

Exclusion Criteria:

* Those with diabetes, incarcerated, bilateral and recurrent hernias and visual problems were excluded from the investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-04; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
postoperative pain using VAS (visual analogue scale) | 1 year

SECONDARY OUTCOMES:
postoperative hyposthesia using VAS (visual analogue scale) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: fatemeh malekpour, MD, Principal Investigator — Shahid Beheshti University of Medical Sciences